CLINICAL TRIAL: NCT03424239
Title: Pilot Study for Zoledronic Acid to Prevent High-Turnover Bone Loss After Bariatric Surgery
Brief Title: Pilot Study for Zoledronic Acid to Prevent Bone Loss After Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elaine W. Yu, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P002081
Record Dates: First submitted 2018-01-23; First posted 2018-02-06 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Bariatric Surgery Candidate
Keywords: Roux-en-Y gastric bypass, sleeve gastrectomy
MeSH Terms: interventions — Zoledronic Acid; Calcium Citrate; Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: All of the participants will receive zoledronic acid, as well as supplementation with calcium and vitamin D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug: Zoledronic Acid, Calcium+Vitamin D (Experimental): Subjects will receive a single intravenous infusion of zoledronic acid (5 mg). Supplemental calcium citrate + vitamin D (500mg+500IU) and vitamin D3 (1000 IU) will be dispensed throughout the study to fit individual needs.
  Interventions: Drug: Zoledronic Acid; Dietary Supplement: Calcium citrate + vitamin D; Dietary Supplement: Vitamin D3

INTERVENTIONS:
Drug: Zoledronic Acid — 5mg zoledronic acid
  Other Names: National Drug Code (NDC) 25021-830-82
Dietary Supplement: Calcium citrate + vitamin D — Chewable 500mg calcium citrate with 500 International Units (IU) Vitamin D3
Dietary Supplement: Vitamin D3 — 1000IU Vitamin D3 gummy

SUMMARY:
This study evaluates whether zoledronic acid can prevent the high bone turnover that occurs after Roux-en-Y Gastric Bypass (RYGB) and sleeve gastrectomy (SG) surgery.

DETAILED DESCRIPTION:
The investigators are evaluating the ability of a single dose of zoledronic acid to improve bone outcomes after RYGB or SG surgery. The investigators have previously shown that RYGB and SG have negative effects on bone density, bone microarchitecture, and that bariatric procedures potentially increase the risk of fractures. The purpose of this study is to evaluate the safety and efficacy of zoledronic acid to prevent the high-turnover bone loss that occurs in adults who have chosen to undergo RYGB or SG.

ELIGIBILITY:
Inclusion Criteria:

* Men must be age ≥ 50
* Women must be age ≥ 25 and postmenopausal
* Planning to receive RYGB or SG surgery

Exclusion Criteria:

* Age < 25
* Prior bariatric surgery
* Weight ≥ 400 lbs
* Liver or renal disease
* Hypercalcemia, hypocalcemia, or hypomagnesemia
* Serum 25-hydroxyvitamin D < 20 ng/mL
* History of bone-modifying disorders
* Use of bone-active medications
* Known sensitivity to bisphosphonates
* Extensive dental work involving extraction or dental implant within the past 2 months or planned in the upcoming 6 months

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine W Yu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: Zoledronic Acid, Calcium+Vitamin D: Subjects will receive a single intravenous infusion of zoledronic acid (5 mg). Supplemental calcium citrate + vitamin D (500mg+500IU) and vitamin D3 (1000 IU) will be dispensed throughout the study to fit individual needs.
  Ergocalciferol 50,000 international units once a day for three days administered prior to Zoledronic Acid
  Zoledronic Acid: 5mg zoledronic acid
  Calcium citrate + vitamin D: Chewable 500mg calcium citrate with 500IU Vitamin D3
  Vitamin D3: 1000IU Vitamin D3 gummy
Period: Overall Study
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
Started | 6
Baseline/Zoledronic Acid Administration | 4
2 Week Post-op | 4
12 Week Post-op | 4
24 Week Post-op | 4
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Drug: Zoledronic Acid, Calcium+Vitamin D: Subjects will receive a single intravenous infusion of zoledronic acid (5 mg). Supplemental calcium citrate + vitamin D (500mg+500IU) and vitamin D3 (1000 IU) will be dispensed throughout the study to fit individual needs.
  Zoledronic Acid: 5mg zoledronic acid
  Calcium citrate + vitamin D: Chewable 500mg calcium citrate with 500IU Vitamin D3
  Vitamin D3: 1000IU Vitamin D3 gummy
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Weight [Mean (Standard Deviation); unit: lb] | 226.0 (18.0)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 40.9 (2.0)
Subtotal body fat [Mean (Standard Deviation); unit: kg] | 46.9 (4.2)
Subtotal body lean mass [Mean (Standard Deviation); unit: kg] | 49.8 (5.8)
Serum calcium [Mean (Standard Deviation); unit: mg/dl] | 9.4 (0.3)
Serum creatinine [Mean (Standard Deviation); unit: mg/dl] | 0.72 (0.14)
Serum 25-hydroxyvitamin D [Mean (Standard Deviation); unit: ng/ml] | 39.8 (14.8)
Serum parathyroid hormone (PTH) [Mean (Standard Deviation); unit: pg/ml] | 43.5 (20.6)
Serum CTX [Mean (Standard Deviation); unit: ng/ml] | 0.226 (0.163)
Serum Procollagen 1 Intact N-Terminal Propeptide (P1NP) [Mean (Standard Deviation); unit: ug/l] | 35.6 (12.5)
DXA Spine areal bone mineral density (aBMD) [Mean (Standard Deviation); unit: g/cm^2] | 1.065 (0.095)
DXA Femoral neck aBMD [Mean (Standard Deviation); unit: g/cm^2] | 0.811 (0.124)
DXA Total hip aBMD [Mean (Standard Deviation); unit: g/cm^2] | 0.953 (0.124)
QCT Trabecular spine volumetric bone mineral density (vBMD) [Mean (Standard Deviation); unit: mg/cm^3] | 114 (41)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum CTX
Description: The primary aim of this study is to determine the postoperative changes in serum markers of bone turnover after a preoperative infusion of zoledronic acid. Serum C-terminal telopeptide of type 1 collagen (CTX) is marker of bone resorption.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
Number analyzed (Participants) | 4
ng/ml | 0.228 (0.117)

2. Secondary Outcome: Change in Total Hip Bone Mineral Density by DXA
Description: Early changes in areal bone mineral density will be measured at the hip and spine by Dual-energy X-ray Absorptiometry (DXA).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
Number analyzed (Participants) | 4
g/cm^2 | -0.039 (0.041)

3. Secondary Outcome: Change in Trabecular Spine Bone Mineral Density by QCT
Description: Early changes in volumetric bone mineral density will be measured at the spine by Quantitative Computed Tomography (QCT).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
Number analyzed (Participants) | 4
mg/cm^3 | 4.9 (7.8)

4. Secondary Outcome: Number of Participants With Treatment-related Hypocalcemia Events as Assessed by CTCAE v4.0
Description: Hypocalcemia, if detected, will be graded according to common terminology for adverse event criteria (CTCAE v.4). Adverse events considered related or possibly related are counted.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
Number analyzed (Participants) | 4
Participants | 0

5. Secondary Outcome: Change From Baseline of Femoral Neck Bone Density Measured by DXA
Description: as for outcome 2
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
Number analyzed (Participants) | 4
g/cm^2 | -0.038 (0.032)

6. Secondary Outcome: Change From Baseline of Spine Bone Density Measured by DXA
Description: as for outcome 2
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
Number analyzed (Participants) | 4
g/cm^2 | 0.003 (0.074)

ADVERSE EVENTS:
Time Frame: 6 to 7 months, starting with pre-surgical drug administration and following until 24 weeks after surgery.
Description: We used definitions consistent with CTCAE version 4.0
Arm/Group | Drug: Zoledronic Acid, Calcium+Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Zoledronic Acid, Calcium+Vitamin D (N=4)
Vertigo (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Zoledronic Acid, Calcium+Vitamin D (N=4)
Fever and body aches (General disorders) | 2 (2)
Diverticulitis flair (Gastrointestinal disorders) | 1 (1)
Post-op GI pain (Gastrointestinal disorders) | 1 (1)
pseudogout flair (Immune system disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT03424239/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT03424239/ICF_002.pdf